CLINICAL TRIAL: NCT05259345
Title: Comparison of Subcostal Exterior Semilunaris Transverses Abdomens, Modified Thoracoabdominal Nerves Block Through Perichondrial Approach, and Rectus Sheath Block in Patients Undergoing Major Abdominal Surgeries
Brief Title: Comparison of SE-TAP, M-TAPA, and Rectus Sheath Block in Abdominal Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gulay ERDOGAN KAYHAN, Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ESOGU anaesthesia
Record Dates: First submitted 2022-02-14; First posted 2022-02-28 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Pain
Keywords: fascial plane blocks; postoperative pain; opioid consumption; quality of recovery; abdominal surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group SE-TAP block (Active Comparator): Bilateral subcostal exterior semilunaris transverses abdominis plane (SE-TAP) block will be performed with 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline)
  Interventions: Procedure: Bilateral SE-TAP
- Group M-TAPA block (Active Comparator): Bilateral modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) will be performed with 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline)
  Interventions: Procedure: Bilateral M-TAPA
- Group RS block (Active Comparator): Bilateral rectus sheath block will be performed with 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline)
  Interventions: Procedure: Bilateral RSB

INTERVENTIONS:
Procedure: Bilateral SE-TAP — A 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline) will be given between the internal oblique and transversus abdominis muscles toward the lateral border of the semilunar along the costal margin.
  Other Names: Ultrasound guided bilateral subcostal exterior semilunaris transversus abdomens plane block
  Arms: Group SE-TAP block
Procedure: Bilateral M-TAPA — A 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline) will be given into the layer between the transverse abdominal muscle and the inferior plane of the costal cartilage at the midclavicular line, in the sagittal plane.
  Other Names: Ultrasound guided bilateral modified thoracoabdominal nerves block through perichondrial approach (M-TAPA)
  Arms: Group M-TAPA block
Procedure: Bilateral RSB — A 20 mL of local anesthetic solution (10 mL of 5% bupivacaine + 5 mL of 2% lidocaine + 5 mL of saline) will be given between the rectus muscle and posterior rectus sheath bilaterally.
  Other Names: Ultrasound guided bilateral rectus sheath block
  Arms: Group RS block

SUMMARY:
The aim of this randomised controlled study is to compare the effects of three different fascial plane block [subcostal exterior semilunaris transverses abdominis plane (SE-TAP) block, modified thoracoabdominal nerves block through perichondrial approach (M-TAPA), and rectus sheath block (RSB)] on postoperative pain levels and opioid consumption in patients undergoing major abdominal surgeries with midline incision.

DETAILED DESCRIPTION:
In last decade,ultrasound guided truncal fascial plane blocks such as transverses abdominis plane (TAP) block and rectus sheath block (RSB) have become popular as a part of postoperative multimodal analgesia for abdominal surgeries as the techniques are simple and the target sites are easily identify. Furthermore, the number of newly defined block techniques is daily increasing like M-TAPA and SE-TAP block.

The rectus sheath block (RSB) is an old technique that suite midline incisions and provides analgesia for somatic pain. The local anesthetic is injected into the space between the posterior wall of the rectus abdominis muscle and its sheath, to block the anterior branches of the thoracoabdominal nerves. It has been suggested that both anterior and lateral branches of the T5-T12 thoracoabdominal nerves are blockade in M-TAPA and SE-TAP blocks. So, they may provide better analgesia and quality of recovery for major abdominal surgeries due to presence of drains. However, the extent of the local anaesthetic diffusion and the dermatomal levels are not clear, and there is no randomised clinical trial about these new techniques, to our knowledge.

Patients and Methods: This is a prospective, randomised, double-blind clinical study; carry out on 120 patients schedule for elective major abdominal surgery with midline incision. While the fascia is closed, 1 g paracetamol and 1 mg/kg tramadol will be administered routinely to all patients for postoperative multimodal analgesia. At the end of surgery, patients will be randomly allocated into three groups (40 patients each); bilateral SE-TAP block in Group S, bilateral RSB in Group R, and bilateral M-TAPA block in Group M will be performed under ultrasound guidance. Patient controlled analgesia with intravenous morphine will be started at the recovery room. Postoperative pain levels, opioid consumption, and quality of recovery will be questioned and recorded at the first postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical classification I-III
* Scheduled for elective laparotomy with a midline incision

Exclusion Criteria:

* Not agree to participate in the study
* Have mental status disorders
* Inability to communicate
* Known bleeding and/or coagulation disorders
* Infection at injection site
* Chronic opioid intake

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | At postoperative 24th hours
  Quality of Recovery-40 (QoR-40), a 40-item questionnaire that provides a global score and subscores across five dimensions; patient support, comfort, emotions, physical independence, and pain (minimum score of 40 and maximum of 200).

SECONDARY OUTCOMES:
Postoperative pain | At postoperative 48 hours (2.,6.,12.,18.,24.,48.hours)
  Numeric rating scale pain from 0 (no pain) to 10 (worst pain).
Opioid consumption | At postoperative 48 hours (2.,6.,12.,18.,24.,48.hours)
  Morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Gulay Erdogan Kayhan, Professor, Principal Investigator — Eskisehir Osmangazi University Faculty of Medicine
Locations (1):
- Eskisehir Osmangazi University Faculty of Medicine, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bakshi SG, Mapari A, Shylasree TS. REctus Sheath block for postoperative analgesia in gynecological ONcology Surgery (RESONS): a randomized-controlled trial. Can J Anaesth. 2016 Dec;63(12):1335-1344. doi: 10.1007/s12630-016-0732-9. Epub 2016 Sep 14. PMID 27638294